CLINICAL TRIAL: NCT00819780
Title: A Randomized, Multicenter, Phase 2 Study to Compare the Efficacy of Panitumumab in Combination With mFOLFOX6 to the Efficacy of Bevacizumab in Combination With mFOLFOX6 in Patients With Previously Untreated, KRAS Wild-Type, Unresectable, Metastatic Colorectal Cancer
Brief Title: PEAK: Panitumumab Plus mFOLFOX6 vs. Bevacizumab Plus mFOLFOX6 for First Line Treatment of Metastatic Colorectal Cancer (mCRC) Patients With Wild-Type Kirsten Rat Sarcoma-2 Virus (KRAS) Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20070509
Record Dates: First submitted 2008-11-06; First posted 2009-01-09 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Colon Cancer; Colorectal Cancer; Rectal Cancer; Metastatic Colorectal Cancer
Keywords: Colon Cancer; Colorectal Cancer; Rectal Cancer; Panitumumab; Vectibix; modified FOLFOX 6; mFOLFOX 6; FOLFOX; Bevacizumab; Avastin; First-Line; metastatic
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms; Neoplasm Metastasis | interventions — Panitumumab; Bevacizumab

ARMS (2):
- Panitumumab Plus mFOLFOX6 (Experimental): Participants received 6 mg/kg panitumumab administered by intravenous (IV) infusion and modified FOLFOX6 (mFOLFOX6) chemotherapy regimen consisting of oxaliplatin (85 mg/m^2), leucovorin (400 mg/m^2) and 5-fluorouracil (5-FU) (2400 mg/m^2) administered on Day 1 of every 14-day cycle until disease progression, unacceptable toxicity, withdrawal of consent, or death.
  Interventions: Drug: Panitumumab; Drug: mFOLFOX6
- Bevacizumab Plus mFOLFOX6 (Active Comparator): Participants received 5 mg/kg bevacizumab administered by IV infusion and the mFOLFOX6 regimen consisting of oxaliplatin (85 mg/m^2), leucovorin (400 mg/m^2), followed by 5-FU (2400 mg/m^2) administered on Day 1 of every 14-day cycle until disease progression, unacceptable toxicity, withdrawal of consent, or death.
  Interventions: Drug: Bevacizumab; Drug: mFOLFOX6

INTERVENTIONS:
Drug: Panitumumab — Panitumumab is a fully human immunoglobulin G (IgG)2 monoclonal antibody antagonist directed against human Epidermal Growth Factor receptor (EGFr).
  Other Names: Vectibix
  Arms: Panitumumab Plus mFOLFOX6
Drug: Bevacizumab — Bevacizumab is a humanized monoclonal IgG1 antibody that is directed against Vascular Endothelial Growth Factor (VEGF).
  Other Names: Avastin
  Arms: Bevacizumab Plus mFOLFOX6
Drug: mFOLFOX6 — mFOLFOX6 regimen is a combination therapy of oxaliplatin (85 mg/m^2) administered as a 2-hour infusion on Day 1; leucovorin (400 mg/m^2) administered as a 2-hour infusion on Day 1; followed by a loading dose of 5-fluorouracil (5-FU; 400 mg/m^2) IV bolus administered over approximately 2 to 4 minutes on Day 1, then 5- FU (2400 mg/m^2) via ambulatory pump administered for a period of 46 to 48 hours.

SUMMARY:
The primary objective of this study is to estimate the treatment effect on progression-free survival (PFS) of panitumumab relative to bevacizumab in combination with mFOLFOX6 chemotherapy as first-line therapy in patients with tumors expressing wild-type KRAS, unresectable mCRC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed adenocarcinoma of the colon or rectum in patients with unresectable metastatic (M1) disease
* Patients with at least 1 uni-dimensionally measurable lesion of at least 10 mm per modified Response Evaluation Criteria in Solid Tumors (RECIST) guidelines
* Wild-type KRAS tumor status confirmed by an Amgen approved central laboratory or an experienced laboratory (local laboratory) per local regulatory guidelines using a validated test method
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* Men or women 18 years of age or older
* Adequate hematologic, renal, hepatic, metabolic, and coagulation function

Exclusion Criteria:

* History of prior or concurrent central nervous system (CNS) metastases
* Prior chemotherapy or other systemic anticancer therapy for treatment of metastatic colorectal carcinoma
* Clinically significant cardiac disease
* Clinically significant peripheral sensory neuropathy
* Active inflammatory bowel disease
* Recent gastroduodenal ulcer to be active or uncontrolled
* History of interstitial lung disease
* Recent pulmonary embolism, deep vein thrombosis, or other significant venous event
* Pre-existing bleeding diathesis and/or coagulopathy with exception of well-controlled anticoagulation therapy
* Recent major surgical procedure, open biopsy, or significant traumatic injury not yet recovered from prior major surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2009-04-24 (Actual); Primary Completion 2012-05-30 (Actual); Study Completion 2016-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (93):
- United States (62):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Berkeley, California
  - Research Site, Beverly Hills, California
  - Research Site, Burbank, California
  - Research Site, Fountain Valley, California
  - Research Site, La Verne, California
  - Research Site, Orange, California
  - Research Site, Riverside, California
  - Research Site, Roseville, California
  - Research Site, Denver, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Boynton Beach, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Alpharetta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Post Falls, Idaho
  - Research Site, Gurnee, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Danville, Kentucky
  - Research Site, Hazard, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Kalamazoo, Michigan
  - Research Site, Lambertville, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Mountain Lakes, New Jersey
  - Research Site, Sparta, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, East Setauket, New York
  - Research Site, Staten Island, New York
  - Research Site, Huntersville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Temple, Texas
  - Research Site, Tyler, Texas
  - Research Site, White River Junction, Vermont
  - Research Site, Chesapeake, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Vancouver, Washington
- Belgium (4):
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Libramont
  - Research Site, Sint-Niklaas
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Oshawa, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Germany (7):
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Magdeburg
  - Research Site, MÃ¼nchen
  - Research Site, Passau
  - Research Site, Regensburg
  - Research Site, WÃ¼rzburg
- Italy (6):
  - Research Site, Alba (CN)
  - Research Site, Fano
  - Research Site, Genova
  - Research Site, Mantova
  - Research Site, Udine
  - Research Site, Varese
- Spain (6):
  - Research Site, MÃ¡laga, AndalucÃ-a
  - Research Site, Santander, Cantabria
  - Research Site, Sabadell, CataluÃ±a
  - Research Site, Elche, Comunidad
  - Research Site, A CoruÃ±a, Galicia
  - Research Site, San SebastiÃ¡n de Los Reyes, Madrid

REFERENCES:
- [Background] Rivera F, Karthaus M, Hecht JR, Sevilla I, Forget F, Fasola G, Canon JL, Guan X, Demonty G, Schwartzberg LS. Final analysis of the randomised PEAK trial: overall survival and tumour responses during first-line treatment with mFOLFOX6 plus either panitumumab or bevacizumab in patients with metastatic colorectal carcinoma. Int J Colorectal Dis. 2017 Aug;32(8):1179-1190. doi: 10.1007/s00384-017-2800-1. Epub 2017 Apr 19. PMID 28424871
- [Background] Schwartzberg LS, Rivera F, Karthaus M, Fasola G, Canon JL, Hecht JR, Yu H, Oliner KS, Go WY. PEAK: a randomized, multicenter phase II study of panitumumab plus modified fluorouracil, leucovorin, and oxaliplatin (mFOLFOX6) or bevacizumab plus mFOLFOX6 in patients with previously untreated, unresectable, wild-type KRAS exon 2 metastatic colorectal cancer. J Clin Oncol. 2014 Jul 20;32(21):2240-7. doi: 10.1200/JCO.2013.53.2473. Epub 2014 Mar 31. PMID 24687833
- [Background] Boeckx N, Koukakis R, Op de Beeck K, Rolfo C, Van Camp G, Siena S, Tabernero J, Douillard JY, Andre T, Peeters M. Primary tumor sidedness has an impact on prognosis and treatment outcome in metastatic colorectal cancer: results from two randomized first-line panitumumab studies. Ann Oncol. 2017 Aug 1;28(8):1862-1868. doi: 10.1093/annonc/mdx119. PMID 28449055
- [Background] Heinemann V, Rivera F, O'Neil BH, Stintzing S, Koukakis R, Terwey JH, Douillard JY. A study-level meta-analysis of efficacy data from head-to-head first-line trials of epidermal growth factor receptor inhibitors versus bevacizumab in patients with RAS wild-type metastatic colorectal cancer. Eur J Cancer. 2016 Nov;67:11-20. doi: 10.1016/j.ejca.2016.07.019. Epub 2016 Sep 1. PMID 27592068
- [Background] Modest DP, Rivera F, Bachet JB, de Braud F, Pietrantonio F, Koukakis R, Demonty G, Douillard JY. Panitumumab-based maintenance after oxaliplatin discontinuation in metastatic colorectal cancer: A retrospective analysis of two randomised trials. Int J Cancer. 2019 Jul 15;145(2):576-585. doi: 10.1002/ijc.32110. Epub 2019 Jan 24. PMID 30614531
- [Background] Peeters M, Forget F, Karthaus M, Valladares-Ayerbes M, Zaniboni A, Demonty G, Guan X, Rivera F. Exploratory pooled analysis evaluating the effect of sequence of biological therapies on overall survival in patients with RAS wild-type metastatic colorectal carcinoma. ESMO Open. 2018 Feb 24;3(2):e000297. doi: 10.1136/esmoopen-2017-000297. eCollection 2018. PMID 29531837
- [Background] Taieb J, Geissler M, Rivera F, Karthaus M, Wilson R, Loupakis F, Price T, Tracy M, Burdon P, Peeters M. Relationship Between Tumor Response and Tumor-Related Symptoms in RAS Wild-Type Metastatic Colorectal Cancer: Retrospective Analyses From 3 Panitumumab Trials. Clin Colorectal Cancer. 2019 Dec;18(4):245-256.e5. doi: 10.1016/j.clcc.2019.07.009. Epub 2019 Jul 29. PMID 31515083
- [Background] Taieb J, Rivera F, Siena S, Karthaus M, Valladares-Ayerbes M, Gallego J, Geissler M, Koukakis R, Demonty G, Peeters M. Exploratory analyses assessing the impact of early tumour shrinkage and depth of response on survival outcomes in patients with RAS wild-type metastatic colorectal cancer receiving treatment in three randomised panitumumab trials. J Cancer Res Clin Oncol. 2018 Feb;144(2):321-335. doi: 10.1007/s00432-017-2534-z. Epub 2017 Oct 28. PMID 29080924
- [Background] Boeckx N, Koukakis R, Op de Beeck K, Rolfo C, Van Camp G, Siena S, Tabernero J, Douillard JY, Andre T, Peeters M. Effect of Primary Tumor Location on Second- or Later-line Treatment Outcomes in Patients With RAS Wild-type Metastatic Colorectal Cancer and All Treatment Lines in Patients With RAS Mutations in Four Randomized Panitumumab Studies. Clin Colorectal Cancer. 2018 Sep;17(3):170-178.e3. doi: 10.1016/j.clcc.2018.03.005. Epub 2018 Mar 8. PMID 29627309
- [Background] Peeters M, Price T, Taieb J, Geissler M, Rivera F, Canon JL, Pentheroudakis G, Koukakis R, Burdon P, Siena S. Relationships between tumour response and primary tumour location, and predictors of long-term survival, in patients with RAS wild-type metastatic colorectal cancer receiving first-line panitumumab therapy: retrospective analyses of the PRIME and PEAK clinical trials. Br J Cancer. 2018 Aug;119(3):303-312. doi: 10.1038/s41416-018-0165-z. Epub 2018 Jul 17. PMID 30013091
- [Background] Sartore-Bianchi A, Garcia-Alfonso P, Geissler M, Kohne CH, Peeters M, Price T, Valladares-Ayerbes M, Zhang Y, Burdon P, Taieb J, Modest DP. Relationships Between Kohne Category/Baseline Tumor Load and Early Tumor Shrinkage, Depth of Response, and Outcomes in Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2021 Dec;20(4):305-313. doi: 10.1016/j.clcc.2021.05.007. Epub 2021 May 25. PMID 34172397
- [Derived] Peeters M, Kafatos G, Taylor A, Gastanaga VM, Oliner KS, Hechmati G, Terwey JH, van Krieken JH. Prevalence of RAS mutations and individual variation patterns among patients with metastatic colorectal cancer: A pooled analysis of randomised controlled trials. Eur J Cancer. 2015 Sep;51(13):1704-13. doi: 10.1016/j.ejca.2015.05.017. Epub 2015 Jun 3. PMID 26049686
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was enrolled on 24 April 2009; last patient was enrolled on 09 December 2011.
Groups:
- Panitumumab Plus mFOLFOX6: Participants received 6 mg/kg panitumumab administered by intravenous (IV) infusion and modified FOLFOX6 (mFOLFOX6) chemotherapy regimen consisting of oxaliplatin (85 mg/m^2), leucovorin (400 mg/m^2) and 5-fluorouracil (5-FU; 2400 mg/m^2) administered on Day 1 of every 14-day cycle until disease progression, unacceptable toxicity, withdrawal of consent, or death.
Period: Overall Study
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Started | 142 | 143
Received Study Treatment | 139 | 139
Completed | 114 (Indicates participants who ended study treatment) | 122 (Indicates participants who ended study treatment)
Not Completed | 28 | 21
Not completed — Did not receive study drug | 3 | 4
Not completed — Still in treatment | 25 | 17

BASELINE CHARACTERISTICS:
Groups:
- Panitumumab Plus mFOLFOX6: Participants received 6 mg/kg panitumumab administered by intravenous (IV) infusion and mFOLFOX6 chemotherapy regimen on Day 1 of every 14-day cycle.
- Bevacizumab Plus mFOLFOX6: Participants received 5 mg/kg bevacizumab administered by IV infusion and the mFOLFOX6 chemotherapy regimen on Day 1 of every 14-day cycle.
- Total: Total of all reporting groups
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6 | Total
Number analyzed (Participants) | 142 | 143 | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.4) | 60.5 (9.8) | 61.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 47 | 103
  Male | 86 | 96 | 182
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 131 | 127 | 258
  Black or African American | 9 | 6 | 15
  Hispanic or Latino | 2 | 5 | 7
  Asian | 0 | 4 | 4
  Japanese | 0 | 1 | 1
Prior Adjuvant Oxaliplatin Therapy [Number; unit: participants]
  Yes | 14 | 14 | 28
  No | 128 | 129 | 257
RAS and BRAF Mutation Status [Number; unit: participants] — This analysis was performed on tumors from 136 and 137 participants in each treatment group respectively. BRAF = v-raf murine sarcoma viral oncogene homolog B1; RAS = rat sarcoma viral oncogene homolog, and includes Kirsten rat sarcoma-2 viral oncogene (KRAS) exons 2, 3 & 4 and neuroblastoma RAS viral (v-ras) oncogene (NRAS) exons 2, 3, and 4. Participants may appear in more than one category.
  participants
    BRAF wild-type | 103 | 108 | 211
    RAS Wild-type | 88 | 82 | 170
    RAS/BRAF wild-type | 77 | 79 | 156
    Testing not performed | 13 | 18 | 31
    Sample acceptance failure | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of first disease progression, or death within 60 days after the last evaluable tumor assessment or randomization date (whichever was later). Participants not meeting the criteria by the cutoff date were censored at the last evaluable tumor assessment date. Tumor response was evaluated by the investigator per modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0 every 8 weeks until radiographic disease progression. Progression is defined as at least a 20% increase in the size of target lesions, unequivocal progression of existing non-target lesions, or any new lesions.
Time Frame: From randomization until the data cutoff date of 30 May 2012; median follow-up time was 60 weeks.
Population: Intent-to-treat (ITT) analysis set (all randomized participants)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 142 | 143
months | 10.9 [9.4 to 13.0] | 10.1 [9.0 to 12.6]
Statistical Analysis 1: Comparison: Panitumumab Plus mFOLFOX6 vs Bevacizumab Plus mFOLFOX6; Test type: Superiority or Other; p = 0.3531, Stratified Cox proportional hazards; The Cox proportional hazard model is stratified by prior adjuvant oxaliplatin therapy; Cox Proportional Hazard = 0.871, 95% CI 2-sided [0.651 to 1.166] — A hazard ratio < 1.0 favors panitumumab

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to the date of death, with participants alive or lost to follow-up at the analysis data cutoff date censored at their last contact date.
Time Frame: From randomization until the data cutoff date of 30 May 2012; median follow-up time was 60 weeks.
Population: Intent-to-treat analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 142 | 143
months | NA [28.8 to NA] — Not estimable due to the low number of events | 25.4 [22.9 to 29.5]
Statistical Analysis 1: Comparison: Panitumumab Plus mFOLFOX6 vs Bevacizumab Plus mFOLFOX6; Test type: Superiority or Other; p = 0.1386, Stratified Cox proportional hazards; The Cox proportional hazard model is stratified by prior adjuvant oxaliplatin therapy; Cox Proportional Hazard = 0.723, 95% CI 2-sided [0.470 to 1.111] — A hazard ratio < 1.0 favors panitumumab

3. Secondary Outcome: Percentage of Participants With an Objective Response
Description: Objective response was defined as having a confirmed complete response (CR) or partial response (PR) during first-line treatment, based on the investigator's review of scans using a modified-RECIST v1.0. A complete or partial response was confirmed no less than 4-weeks after the criteria for response were first met. Complete Response: Disappearance of all target and non-target lesions and no new lesions. Partial Response: At least a 30% decrease in the sum of the longest diameter (SLD) of target lesions and no progression of non-target lesions and no new lesions, or the disappearance of all target lesions with persistence of one or more non-target lesion(s) not qualifying for either CR or progressive disease and no new lesions.
Time Frame: From randomization until the data cutoff date of 30 May 2012; median follow-up time was 60 weeks.
Population: Evaluable for Local Tumor Response Analysis Set, defined as the subset of participants in the ITT Analysis Set who had at least 1 unidimensionally measurable lesion per modified RECIST 1.0 per the local investigator.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 142 | 142
percentage of participants | 57.75 [49.18 to 65.98] | 53.52 [44.97 to 61.93]
Statistical Analysis 1: Comparison: Panitumumab Plus mFOLFOX6 vs Bevacizumab Plus mFOLFOX6; Test type: Superiority or Other; p = 0.5497, Stratified exact test; Stratified by prior adjuvant oxaliplatin therapy; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.72 to 1.95] — The odds ratio is defined as the odds of having an objective response in the panitumumab plus mFOLFOX6 arm relative to the odds in the bevacizumab plus mFOLFOX6 arm

4. Secondary Outcome: Duration of Response
Description: For participants with a confirmed objective response, the time from first confirmed objective response to radiologic disease progression per modified RECIST 1.0 criteria or death. For participants who responded and have not progressed or died, duration of response was censored at their last evaluable disease assessment date.
Time Frame: From randomization until the data cutoff date of 30 May 2012; median follow-up time was 60 weeks.
Population: Evaluable for Local Tumor Response Analysis Set: Responders
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 82 | 76
months | 10.0 [8.4 to 12.9] | 9.0 [7.4 to 9.5]

5. Secondary Outcome: Time to Disease Progression
Description: Time to progression (TTP) is defined as the time from randomization to the date of radiologic disease progression per modified RECIST 1.0 criteria. Participants not meeting criteria for disease progression by the analysis data cutoff date were censored at their last evaluable disease assessment date. Progression is defined as at least a 20% increase in the size of target lesions, unequivocal progression of existing non-target lesions, or any new lesions.
Time Frame: From randomization until the data cutoff date of 30 May 2012; median follow-up time was 60 weeks.
Population: Intent-to-treat analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 142 | 143
months | 11.0 [9.7 to 13.1] | 11.1 [9.3 to 12.7]
Statistical Analysis 1: Comparison: Panitumumab Plus mFOLFOX6 vs Bevacizumab Plus mFOLFOX6; Test type: Superiority or Other; p = 0.3861, Stratified Cox proportional hazards; The Cox proportional hazard model is stratified by prior adjuvant oxaliplatin therapy; Cox Proportional Hazard = 0.874, 95% CI 2-sided [0.645 to 1.185] — A hazard ratio < 1.0 favors panitumumab

6. Secondary Outcome: Time to Initial Objective Response
Description: For participants with a confirmed objective response, the time from randomization to the date of first confirmed objective response. Assessments are based on the investigator's review of scans using a modified-RECIST v1.0. An objective response is defined as a best tumor response of complete or partial response. A complete or partial response was confirmed no less than 4-weeks after the criteria for response were first met.
Time Frame: From randomization until the data cutoff date of 30 May 2012; median follow-up time was 60 weeks.
Population: Evaluable for Local Tumor Response Analysis Set: Responders
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 82 | 76
months | 1.8 [1.7 to 2.3] | 1.9 [1.7 to 3.7]

7. Secondary Outcome: Resection Rate
Description: The resection rate was defined as the percentage of participants with a surgical procedure that resulted in partial reduction or complete eradication of all metastatic disease.
Time Frame: From randomization until the data cutoff date of 30 May 2012; median follow-up time was 60 weeks.
Population: Intent-to-treat analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 142 | 143
percentage of participants | 12.68 [7.69 to 19.29] | 11.19 [6.53 to 17.53]

8. Secondary Outcome: Progression-free Survival (PFS) in Participants With Wild-type Rat Sarcoma Viral Oncogene Homolog (RAS)
Description: as for outcome 1
Time Frame: From randomization until the data cutoff date of 30 May 2012; median follow-up time was 60 weeks.
Population: Wild-type RAS Efficacy Analysis Set, defined as a subset of Wild-type KRAS Exon 2 Efficacy Analysis Set including all randomized participants with wild-type KRAS exon 2, 3, 4, NRAS exon 2, 3, and 4.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 88 | 82
months | 13.0 [10.9 to 15.1] | 9.5 [9.0 to 12.7]
Statistical Analysis 1: Comparison: Panitumumab Plus mFOLFOX6 vs Bevacizumab Plus mFOLFOX6; Test type: Superiority or Other; p = 0.0286, Stratified Cox proportional hazards; The Cox proportional hazard model is stratified by prior adjuvant oxaliplatin therapy; Cox Proportional Hazard = 0.651, 95% CI 2-sided [0.444 to 0.956] — A hazard ratio < 1.0 favors panitumumab

9. Secondary Outcome: Progression-free Survival (PFS) in Participants With Wild-type RAS / V-raf Murine Sarcoma Viral Oncogene Homolog B1 (BRAF)
Description: as for outcome 1
Time Frame: From randomization until the data cutoff date of 30 May 2012; median follow-up time was 60 weeks.
Population: Wild-type RAS/BRAF Efficacy Analysis Set was defined as a subset of Wild-type KRAS Exon 2 Efficacy Analysis Set with wild-type KRAS exon 2, 3, and 4, NRAS exon 2, 3, 4, and BRAF exon 15.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 77 | 79
months | 13.1 [10.9 to 15.8] | 9.7 [7.9 to 12.7]
Statistical Analysis 1: Comparison: Panitumumab Plus mFOLFOX6 vs Bevacizumab Plus mFOLFOX6; Test type: Superiority or Other; p = 0.0083, Stratified Cox proportional hazards; The Cox proportional hazard model is stratified by prior adjuvant oxaliplatin therapy; Cox Proportional Hazard = 0.579, 95% CI 2-sided [0.386 to 0.869] — A hazard ratio < 1.0 favors panitumumab

10. Secondary Outcome: Overall Survival in Participants With Wild-type RAS
Description: as for outcome 2
Time Frame: From randomization until the data cutoff date of 30 May 2012; median follow-up time was 60 weeks.
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 88 | 82
months | NA [28.8 to NA] — Could not be estimated due to the low number of events | 29.0 [24.3 to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Panitumumab Plus mFOLFOX6 vs Bevacizumab Plus mFOLFOX6; Test type: Superiority or Other; p = 0.0934, Stratified Cox proportional hazards; The Cox proportional hazard model is stratified by prior adjuvant Oxaliplatin therapy; Cox Proportional Hazard = 0.606, 95% CI 2-sided [0.337 to 1.088] — A hazard ratio < 1.0 favors panitumumab

11. Secondary Outcome: Overall Survival in Participants With Wild-type RAS / BRAF
Description: as for outcome 2
Time Frame: From randomization until the data cutoff date of 30 May 2012; median follow-up time was 60 weeks.
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 77 | 79
months | NA [NA to NA] — Could not be estimated due to the low number of events | 29.0 [24.3 to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Panitumumab Plus mFOLFOX6 vs Bevacizumab Plus mFOLFOX6; Test type: Superiority or Other; p = 0.0235, Stratified Cox proportional hazards; The Cox proportional hazard model is stratified by prior adjuvant oxaliplatin therapy; Cox Proportional Hazard = 0.465, 95% CI 2-sided [0.239 to 0.902] — A hazard ratio < 1.0 favors panitumumab

12. Secondary Outcome: Percentage of Participants With an Objective Response for Participants With Wild-type RAS
Description: as for outcome 3
Time Frame: From randomization until the data cutoff date of 30 May 2012; median follow-up time was 60 weeks.
Population: Wild-type RAS Investigator Tumor Response Analysis Set, defined as the subset of participants in the Wild-type RAS Efficacy Analysis Set who had at least 1 unidimensionally measurable lesion per modified RECIST 1.0 per the local investigator.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 88 | 81
percentage of participants | 63.64 [52.69 to 73.63] | 60.49 [49.01 to 71.19]
Statistical Analysis 1: Comparison: Panitumumab Plus mFOLFOX6 vs Bevacizumab Plus mFOLFOX6; Test type: Superiority or Other; p = 0.9426, Stratified exact test; Stratified by prior exposure to oxaliplatin; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.55 to 2.12] — [estimate comment as in outcome 3, analysis 1]

13. Secondary Outcome: Percentage of Participants With an Objective Response for Participants With Wild-type RAS / BRAF
Description: as for outcome 3
Time Frame: From randomization until the data cutoff date of 30 May 2012; median follow-up time was 60 weeks.
Population: Wild-type RAS/BRAF Investigator Tumor Response Analysis Set, defined as the subset of participants in the Wild-type RAS/BRAF Efficacy Analysis Set who had at least 1 unidimensionally measurable lesion per modified RECIST 1.0 per the local investigator.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 77 | 78
percentage of participants | 63.64 [51.88 to 74.30] | 61.54 [49.83 to 72.34]
Statistical Analysis 1: Comparison: Panitumumab Plus mFOLFOX6 vs Bevacizumab Plus mFOLFOX6; Test type: Superiority or Other; p = 1.0000, Stratified exact test; Stratified by prior exposure to oxaliplatin; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.52 to 2.15] — [estimate comment as in outcome 3, analysis 1]

14. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Severity was graded using Common Terminology Criteria for Adverse Events (CTCAE) v3.0, with the exception of some dermatology/skin adverse events that were graded using CTCAE v3.0 with modifications. Fatal adverse events are classified as grade 5. Serious adverse events include any event that is fatal, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or other significant medical hazard. Treatment-related AEs were those that the investigator considered a reasonable possibility that might have been caused by study drug.
Time Frame: The time frame for adverse event reporting is from the first dose date to 30 days since the last dose date. The median time frame is 8.0 months for Panitumumab Plus mFOLFOX arm and 7.3 months for Bevacizumab Plus mFOLFOX6 arm.
Population: Safety analysis set, which included all randomized participants who received at least 1 dose of protocol treatment (ie, panitumumab, bevacizumab, or any component of mFOLFOX6).
Measure: Number; unit: participants
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Number analyzed (Participants) | 139 | 139
participants
  Any adverse event (AE) | 139 | 139
  AE with worst grade of 3 | 88 | 78
  AE with worst grade of 4 | 31 | 28
  AE with worst grade of 5 | 7 | 9
  Serious adverse event (SAE) | 61 | 53
  AE leading to discontinuation of study drug | 34 | 37
  Any treatment-related adverse event (TRAE) | 138 | 136
  Treatment-related AE with worst grade of 3 | 92 | 77
  Treatment-related AE with worst grade of 4 | 24 | 25
  Treatment-related AE with worst grade of 5 | 3 | 2
  Serious treatment-related adverse event | 37 | 28
  TRAE leading to discontinuation of study drug | 28 | 29

ADVERSE EVENTS:
Time Frame: The time frame for adverse event reporting is from the first dose date to 30 days since the last dose date. The median time frame is 8.0 months for Panitumumab Plus Chemotherapy arm and 7.3 months for Bevacizumab Plus Chemotherapy arm.
Description: The table of Other Adverse Events summarizes non-serious occurrences of adverse events that exceeded a 5% frequency in either treatment arm.
Arm/Group | Panitumumab Plus mFOLFOX6 | Bevacizumab Plus mFOLFOX6
Serious Adverse Events (participants affected / at risk) | 61/139 | 53/139
Other Adverse Events (participants affected / at risk) | 139/139 | 139/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus mFOLFOX6 (N=139) | Bevacizumab Plus mFOLFOX6 (N=139)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Anal fistula (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 3
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Intestinal perforation (Gastrointestinal disorders) | 0 | 2
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Rectal perforation (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Adverse drug reaction (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 2 | 4
Thrombosis in device (General disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Herpes zoster oticus (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 2
Infusion site infection (Infections and infestations) | 1 | 0
Meningoencephalitis herpetic (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3
Postoperative wound infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 4
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Substance abuse (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 4
Intra-abdominal haematoma (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus mFOLFOX6 (N=139) | Bevacizumab Plus mFOLFOX6 (N=139)
Anaemia (Blood and lymphatic system disorders) | 24 | 20
Leukopenia (Blood and lymphatic system disorders) | 10 | 9
Neutropenia (Blood and lymphatic system disorders) | 63 | 66
Thrombocytopenia (Blood and lymphatic system disorders) | 34 | 17
Conjunctivitis (Eye disorders) | 16 | 4
Lacrimation increased (Eye disorders) | 7 | 6
Vision blurred (Eye disorders) | 8 | 3
Abdominal pain (Gastrointestinal disorders) | 25 | 25
Abdominal pain upper (Gastrointestinal disorders) | 11 | 12
Cheilitis (Gastrointestinal disorders) | 8 | 0
Constipation (Gastrointestinal disorders) | 44 | 44
Diarrhoea (Gastrointestinal disorders) | 84 | 84
Dyspepsia (Gastrointestinal disorders) | 14 | 15
Flatulence (Gastrointestinal disorders) | 10 | 6
Haemorrhoids (Gastrointestinal disorders) | 4 | 7
Nausea (Gastrointestinal disorders) | 75 | 83
Rectal haemorrhage (Gastrointestinal disorders) | 7 | 6
Stomatitis (Gastrointestinal disorders) | 46 | 31
Vomiting (Gastrointestinal disorders) | 43 | 38
Asthenia (General disorders) | 50 | 44
Chills (General disorders) | 11 | 12
Fatigue (General disorders) | 50 | 65
Mucosal inflammation (General disorders) | 49 | 21
Oedema peripheral (General disorders) | 18 | 13
Pyrexia (General disorders) | 21 | 30
Temperature intolerance (General disorders) | 7 | 11
Bronchitis (Infections and infestations) | 4 | 8
Nasopharyngitis (Infections and infestations) | 7 | 8
Paronychia (Infections and infestations) | 25 | 2
Respiratory tract infection (Infections and infestations) | 7 | 5
Rhinitis (Infections and infestations) | 9 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 9
Urinary tract infection (Infections and infestations) | 9 | 10
Infusion related reaction (Injury, poisoning and procedural complications) | 9 | 6
Platelet count decreased (Investigations) | 10 | 5
Weight decreased (Investigations) | 31 | 16
Weight increased (Investigations) | 8 | 2
Decreased appetite (Metabolism and nutrition disorders) | 56 | 44
Dehydration (Metabolism and nutrition disorders) | 18 | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 12 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 38 | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 57 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 14
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 18
Dizziness (Nervous system disorders) | 16 | 15
Dysaesthesia (Nervous system disorders) | 13 | 23
Dysgeusia (Nervous system disorders) | 31 | 27
Headache (Nervous system disorders) | 12 | 15
Neuropathy peripheral (Nervous system disorders) | 44 | 45
Neurotoxicity (Nervous system disorders) | 15 | 13
Paraesthesia (Nervous system disorders) | 25 | 31
Peripheral sensory neuropathy (Nervous system disorders) | 24 | 24
Polyneuropathy (Nervous system disorders) | 18 | 16
Anxiety (Psychiatric disorders) | 10 | 8
Insomnia (Psychiatric disorders) | 14 | 19
Proteinuria (Renal and urinary disorders) | 15 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 29 | 32
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 12
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 13
Acne (Skin and subcutaneous tissue disorders) | 35 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 21
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 27 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 53 | 12
Erythema (Skin and subcutaneous tissue disorders) | 11 | 2
Exfoliative rash (Skin and subcutaneous tissue disorders) | 11 | 2
Hypertrichosis (Skin and subcutaneous tissue disorders) | 9 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 12 | 6
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 22 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 4
Rash (Skin and subcutaneous tissue disorders) | 86 | 9
Skin fissures (Skin and subcutaneous tissue disorders) | 29 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 8 | 0
Deep vein thrombosis (Vascular disorders) | 5 | 10
Haematoma (Vascular disorders) | 1 | 7
Hypertension (Vascular disorders) | 6 | 35
Hypotension (Vascular disorders) | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.